CLINICAL TRIAL: NCT02748915
Title: Estimation of Perceptual Levels Used in Cochlear Implant Fitting Based on Electrophysiological Measures
Brief Title: Electrophysiological-based Estimation of Cochlear Implant Fitting
Acronym: ENPICME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL15_0309
Record Dates: First submitted 2016-04-14; First posted 2016-04-22 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cochlear Implants
Keywords: Cochlear Implant; ECAP; EABR; perceptual levels; hearing performances

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients using cochlear implants (Experimental): All patients using cochlear implants included in the study will take electrophysiological and psychoacoustic tests to measure auditive parameters regarding the study objectives : ECAP, EABR, speech recognition and MCL.
  Interventions: Other: Electrophysiological and psychoacoustic tests
- Patients using EAS device (Experimental): Patients using EAS device for more than 11 months will take electrophysiological and psychoacoustic tests with the implant functioning only with electrical pulses or in bimodal mode to measure ECAP, EABR, speech recognition and MCL ; this will allow to perform bimodal comparison.
  Interventions: Other: Electrophysiological and psychoacoustic tests
- Patients with bilateral cochlear implant (Experimental): Patients with bilateral cochlear implant for more than 11 months will take electrophysiological and psychoacoustic tests to measure ECAP, EABR, speech recognition, and MCL. The binaural interaction component will also be measured ; this will allow to perform binaural comparison.
  Interventions: Other: Electrophysiological and psychoacoustic tests

INTERVENTIONS:
Other: Electrophysiological and psychoacoustic tests

SUMMARY:
The primary objective of this research is to evaluate the relationships between multiple data from cochlear implant (CI) adult users to and to estimate predictive models of their fitting parameters. In a group of patients, the Electrically-evoked Compound Action Potentials (ECAP) will be collected intra-operatively and the correlation with demographic data (deafness duration, age deafness onset, etiology, duration of cochlear implant use of CI), auditory performances and subjective measures used for implant fitting (hearing threshold and most comfortable level) will be calculated. In a second group of experienced users (more than 9months of use of their CI), ECAP and Electrically-evoked Auditory Brainstem Response (EABR) will be collected after 9 months of CI experience and after 12 months or more of use. Correlation analyzes with demographic data, performance and fitting parameters will be performed as well. Statistical predictive models for both fitting at the activation or in experienced users should be developed according to the correlation analysis.

The secondary objective is to evaluate the effects of simultaneous stimulation on hearing performances. Simultaneous stimulations will be delivered in one ear (bimodal condition) in patients using an Electro-Acoustic Stimulation device (EAS) or in the two ears (binaural condition) for bilateral CI users. ECAP, EABR and speech perception will be measured and compared in the different conditions.

ELIGIBILITY:
Inclusion Criteria:

* Good general health status including no neuropsychological diseases affecting intellectual capacities
* Users of cochlear implant or electro-acoustic stimulation devices
* Normal otoscopy
* No excessive sound exposure within 48h before the measure

Exclusion Criteria:

* For women, possibility of pregnancy (absence of effective contraception or confirmed menopause);
* Concomitant use of ototoxic or psychotropic treatment with anxiolytic and / or antipsychotic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
ECAP threshold | from 11 months after cochlear implant activation
  ECAP amplitude growth function (AGF) will be recorded on three cochlear sites (basal, medial, apical) in all patients using their implants for more than 11 months. ECAP thresholds (in current unit) will be determined, compared according to the stimulation sites and correlation tests with the other measures will be performed. These records could also be compared to ECAP AGF recorded in clinical routine/during control visit before these 11 months that includes intra-operative records when available.
  The ECAP threshold recorded with and without acoustic stimulations will be compared in patients using EAS devices.

SECONDARY OUTCOMES:
ECAP threshold | 9 months after cochlear implant activation
  ECAP AGF will be recorded on three cochlear sites (basal, medial, apical) in all patients using their implants for 9 months. ECAP thresholds (in current unit) will be determined, compared according to the stimulation sites and correlation tests with the other measures will be performed.
ECAP maximal amplitude | from 11 months after cochlear implant activation
  ECAP AGF will be recorded on three cochlear sites (basal, medial, apical) in all patients using their implants for more than 11 months. ECAP maximal amplitudes (in µV) will be determined, compared according to the stimulation sites and correlation tests with the other measures will be performed. These records could also be compared to ECAP AGF recorded in clinical routine/during control visit before these 11 months that includes intra-operative records when available.
  The ECAP amplitude recorded with and without acoustic stimulations will be compared in patients using EAS devices.
ECAP maximal amplitude | 9 months after cochlear implant activation
  ECAP AGF will be recorded on three cochlear sites (basal, medial, apical) in all patients using their implants for 9 months. ECAP maximal amplitudes (in µV) will be determined, compared according to the stimulation sites and correlation tests with the other measures will be performed.
ECAP latency | from 11 months after cochlear implant activation
  ECAP AGF will be recorded on three cochlear sites (basal, medial, apical) in all patients using their implants for more than 11 months. ECAP latencies (in µs) of the ECAP recorded with the highest stimulation level will be determine , compared according to the stimulation sites and correlation tests with the other measures will be performed. These records could also be compared to ECAP AGF recorded in clinical routine/during control visit before these 11 months that includes intra-operative records when available.
  The ECAP latencies recorded with and without acoustic stimulations will be compared in patients using EAS devices.
ECAP latency | 9 months after cochlear implant activation
  ECAP AGF will be recorded on three cochlear sites (basal, medial, apical) in all patients using their implants for 9 months. ECAP latencies (in µs) of the ECAP recorded with the highest stimulation level will be determined, compared according to the stimulation sites and correlation tests with the other measures will be performed.
ECAP AGF slope | from 11 months after cochlear implant activation
  ECAP AGF will be recorded on three cochlear sites (basal, medial, apical) in all patients using their implants for more than 11 months. ECAP AGF slopes (µV/qu) will be determined, compared according to the stimulation sites and correlation tests with the other measures will be performed. These records could also be compared to ECAP AGF recorded in clinical routine/during control visit before these 11 months that includes intra-operative records when available.
  The ECAP AGF slopes recorded with and without acoustic stimulations will be compared in patients using EAS devices.
ECAP AGF slope | 9 months after cochlear implant activation
  ECAP AGF will be recorded on three cochlear sites (basal, medial, apical) in all patients using their implants for 9 months. ECAP AGF slopes (µV/qu) will be determined, compared according to the stimulation sites and correlation tests with the other measures will be performed.
EABR wave V maximal amplitude | from 11 months after cochlear implant activation
  EABR AGF will be recorded on three cochlear sites (basal, medial, apical) in all patients using their implants for more than 11 months. EABR wave V maximal amplitudes (µV) will be determined, compared according to the stimulation sites and correlation tests with the other measures will be performed. These records could also be compared to EABR AGF recorded in clinical routine/during control visit before these 11 months.
EABR wave V maximal amplitude | 9 months after cochlear implant activation
  EABR AGF will be recorded on three cochlear sites (basal, medial, apical) in all patients using their implants for 9 months. EABR wave V maximal amplitudes (µV) will be determined, compared according to the stimulation sites and correlation tests with the other measures will be performed.
EABR wave V latency | from 11 months after cochlear implant activation
  EABR AGF will be recorded on three cochlear sites (basal, medial, apical) in all patients using their implants for more than 11 months. EABR wave V latencies (ms) recorded with the highest stimulation level will be determined, compared according to the stimulation sites and correlation tests with the other measures will be performed. These records could also be compared to EABR AGF recorded in clinical routine/during control visit before these 11 months.
EABR wave V latency | 9 months after cochlear implant activation
  EABR AGF will be recorded on three cochlear sites (basal, medial, apical) in all patients using their implants for 9 months. EABR wave V latencies (ms) recorded with the highest stimulation level will be determined, compared according to the stimulation sites and correlation tests with the other measures will be performed.
EABR wave V threshold | from 11 months after cochlear implant activation
  EABR AGF will be recorded on three cochlear sites (basal, medial, apical) in all patients using their implants for more than 11 months. EABR wave V thresholds (current unit) will be determined, compared according to the stimulation sites and correlation tests with the other measures will be performed. These records could also be compared to EABR AGF recorded in clinical routine/during control visit before these 11 months.
EABR wave V threshold | 9 months after cochlear implant activation
  EABR AGF will be recorded on three cochlear sites (basal, medial, apical) in all patients using their implants for 9 months. EABR wave V thresholds (current unit) will be determined, compared according to the stimulation sites and correlation tests with the other measures will be performed.
EABR wave V AGF slope | from 11 months after cochlear implant activation
  EABR AGF will be recorded on three cochlear sites (basal, medial, apical) in all patients using their implants for more than 11 months. EABR wave V AGF slopes (µV/qu) will be determined, compared according to the stimulation sites and correlation tests with the other measures will be performed. These records could also be compared to EABR AGF recorded in clinical routine/during control visit before these 11 months.
EABR wave V AGF slope | 9 months after cochlear implant activation
  EABR AGF will be recorded on three cochlear sites (basal, medial, apical) in all patients using their implants for 9 months. EABR wave V AGF slopes (µV/qu) will be determined, compared according to the stimulation sites and correlation tests with the other measures will be performed.
EABR binaural interaction component (BIC) | from 11 months after cochlear implant activation
  In bilaterally implanted patients using both of their implants for more than 11 months, EABR BIC will be recorded with a reference electrode of either the older implant or the one associated with the best hearing performances and all the electrodes of the second implant. EABR BIC amplitude (µV) will be determined, compared according to the electrode pairing and correlation tests with the other measures will be performed.
Most Comfort Level (MCL) | from 11 months after cochlear implant activation
  The MCL (current unit) will be evaluated for each electrode/cochlear site tested during the same recording session than the ECAP threshold evaluated after 11 months. These subjective limits will be compared according to the stimulation sites and correlated to ECAP and/or EABR characteristics.
Most Comfort Level (MCL) | 9 months after implant cochlear implant activation
  The MCL (current unit) will be evaluated for each electrode/cochlear site tested during the same recording session than the ECAP threshold evaluated at 9 months. These subjective limits will be compared according to the stimulation sites and correlated to ECAP and/or EABR characteristics.
Speech recognition score | from 11 months after implant cochlear implant activation
  The percentage of speech recognition will be measured at 60 decibels (dB) in open space with implant(s) well fitted during the same recording session than the ECAP threshold evaluated after 11 months. This performance level will be correlated to the ECAP and/or EABR characteristics. In the bimodal and binaural groups, performances will be compared between hearing conditions (monaural = 1 implant vs. bimodal or binaural hearing).
  During these audiometry tests, the recognition score will be also measured at 40 and 50 dB and a pure tone audiometry will be performed.
Speech recognition score | 9 months after implant cochlear implant activation
  The percentage of speech recognition will be measured at 60 dB in open space with implant(s) well fitted during the same recording session than the ECAP threshold evaluated at 9 months. This performance level will be correlated to the ECAP and/or EABR characteristics.
  During these audiometry tests, the recognition score will be also measured at 40 and 50 dB and a pure tone audiometry will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Eric TRUY, Professor, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Edouard Herriot - Service ORL Pavillon U, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Joly CA, Reynard P, Hermann R, Seldran F, Gallego S, Idriss S, Thai-Van H. Intra-Cochlear Current Spread Correlates with Speech Perception in Experienced Adult Cochlear Implant Users. J Clin Med. 2021 Dec 13;10(24):5819. doi: 10.3390/jcm10245819. PMID 34945115
- [Result] Joly CA, Pean V, Hermann R, Seldran F, Thai-Van H, Truy E. Using Electrically-evoked Compound Action Potentials to Estimate Perceptive Levels in Experienced Adult Cochlear Implant Users. Otol Neurotol. 2017 Oct;38(9):1278-1289. doi: 10.1097/MAO.0000000000001548. PMID 28834942